CLINICAL TRIAL: NCT04780659
Title: Immunological Responses After Vaccination for COVID-19 With the Messenger Ribonucleic Acid (mRNA) Vaccine Comirnaty in Immunosuppressed and Immunocompetent Individuals. An Open and Non-randomized, Phase IV Multicenter Study
Brief Title: COVID-19 Vaccination of Immunodeficient Persons (COVAXID)
Acronym: COVAXID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Soo Aleman, MD, PhD, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021-000175-37
Record Dates: First submitted 2021-02-19; First posted 2021-03-03 (Actual); Results first posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine; mRNA Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vaccination with Comirnaty according to standard of care treatment (Experimental): All study participants will receive Comirnaty according to current approval.
  Interventions: Biological: Comirnaty (COVID-19, mRNA vaccine)

INTERVENTIONS:
Biological: Comirnaty (COVID-19, mRNA vaccine) — Comirnaty will be administered two times, one at Day 0 and the second dose at Day 21.
  Other Names: tozinameran; Pfizer mRNA vaccine

SUMMARY:
The study is designed as an open, non-randomized, phase IV cohort study in which the mRNA vaccine Comirnaty will be given in two doses. Analyses will be performed on blood and saliva, investigating humoral and cellular vaccine responses. Occurence of local or systemic reactogenicity will be evaluated, as well as adverse events. The study will include persons with primary or secondary immunosuppressive disorders, as well as immunocompetent persons, with the aim of investigating if the immune responses after given Comirnaty mRNA vaccine against COVID-19.

DETAILED DESCRIPTION:
In this study with 450 patients with primary or secondary immunosuppressive disorders (patients with primary immunodeficiency, HIV infected patients, patients with allogenic stem cell transplantation/CAR T cell treated, solid organ transplanted, and patients with chronic lymphatic leukemia) from Karolinska University Hospital, and healthy controls of 90 individuals for comparison, we will investigate the safety and the immune responses after mRNA vaccination with Comirnaty after two doses, under 6 months of time for each participant. The study is In collaboration with research groups at Karolinska Institutet and SciLifeLab, with planned in-depth detailed analyses of antibody responses as well as cellular responses. The study has obtained permission from Swedish Medical Agency and Swedish Ethical Review Authority.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals ≥18 years old

2a. In the opinion of the investigator, individuals with immunosuppressive disease who meet one of the following criteria:

* Primary immunodeficiency
* Human immunodeficiency virus (HIV)-infection
* Allogeneic stem cell transplantation / Chimeric antigen receptor (CAR T cell) therapy
* Solid organ transplant
* Chronic lymphatic leukemia

or

2b. In the opinion of the investigator, individuals without immunosuppressive disease or treatment without significant co-morbidity

3. Provision of signed informed consent to participate in the study

Exclusion Criteria:

1. Previous or ongoing Coronavirus Disease-19 (COVID-19).
2. Coagulation disorders, other conditions associated with prolonged bleeding time or anticoagulant treatments, which according to the investigator contraindicate intramuscular injection. Conditions which can be corrected with measures such as platelet concentrate treatments, coagulation factors or other measures for people responsible for anticoagulants are not exclusion criteria.
3. Planned to receive another vaccine within 14 days before the first dose of the study vaccine, or during the period from the first dose of the study vaccine up to 14 days after the second dose of the study vaccine, and vaccination with another vaccine which in the investigator's opinion cannot be planned outside these time periods
4. Pregnancy or breast feeding.
5. Hypersensitivity to the active substance or to any of the excipients contained in the vaccine
6. Individuals who cannot understand the informed consent.
7. Individuals who for other reasons are considered by investigators as not suitable for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 539 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2024-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Soo Aleman, MD, PhD, Principal Investigator — Karolinska University Hospital, ME Infectious Diseases
Locations (1):
- Karolinska University Hospital, Stockholm, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Will submit data to European Union Drug Regulating Authorities Clinical Trials Database (EudraCT) and share data result. Will share research results and data through national COVID-19 data portal, operated by SciLifeLab Data Centre, Sweden.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Within one year after study end.
Access Criteria: Published in EudraCT and national COVID-19 data portal (SciLifeLab Data Centre)
URL: https://eudract.ema.europa.eu/index.html

REFERENCES:
- [Derived] Chen P, Bergman P, Blennow O, Hansson L, Mielke S, Nowak P, Gao Y, Soderdahl G, Osterborg A, Smith CIE, Vesterbacka J, Wullimann D, Cuapio A, Akber M, Bogdanovic G, Muschiol S, Aberg M, Lore K, Chen MS, Ljungman P, Buggert M, Aleman S, Ljunggren HG. Real-world assessment of immunogenicity in immunocompromised individuals following SARS-CoV-2 mRNA vaccination: a two-year follow-up of the prospective clinical trial COVAXID. EBioMedicine. 2024 Nov;109:105385. doi: 10.1016/j.ebiom.2024.105385. Epub 2024 Oct 11. PMID 39395230
- [Derived] Chen P, Bergman P, Blennow O, Hansson L, Mielke S, Nowak P, Soderdahl G, Osterborg A, Smith CIE, Vesterbacka J, Wullimann D, Cuapio A, Akber M, Bogdanovic G, Muschiol S, Aberg M, Lore K, Sallberg Chen M, Buggert M, Ljungman P, Aleman S, Ljunggren HG. Real-world assessment of immunogenicity in immunocompromised individuals following SARS-CoV-2 mRNA vaccination: a one-year follow-up of the prospective clinical trial COVAXID. EBioMedicine. 2023 Aug;94:104700. doi: 10.1016/j.ebiom.2023.104700. Epub 2023 Jul 13. PMID 37453361
- [Derived] Cuapio A, Boulouis C, Filipovic I, Wullimann D, Kammann T, Parrot T, Chen P, Akber M, Gao Y, Hammer Q, Strunz B, Perez Potti A, Rivera Ballesteros O, Lange J, Muvva JR, Bergman P, Blennow O, Hansson L, Mielke S, Nowak P, Soderdahl G, Osterborg A, Smith CIE, Bogdanovic G, Muschiol S, Hellgren F, Lore K, Sobkowiak MJ, Gabarrini G, Healy K, Sallberg Chen M, Alici E, Bjorkstrom NK, Buggert M, Ljungman P, Sandberg JK, Aleman S, Ljunggren HG. NK cell frequencies, function and correlates to vaccine outcome in BNT162b2 mRNA anti-SARS-CoV-2 vaccinated healthy and immunocompromised individuals. Mol Med. 2022 Feb 8;28(1):20. doi: 10.1186/s10020-022-00443-2. PMID 35135470
- [Derived] Healy K, Pin E, Chen P, Soderdahl G, Nowak P, Mielke S, Hansson L, Bergman P, Smith CIE, Ljungman P, Valentini D, Blennow O, Osterborg A, Gabarrini G, Al-Manei K, Alkharaan H, Sobkowiak MJ, Yousef J, Mravinacova S, Cuapio A, Xu X, Akber M, Lore K, Hellstrom C, Muschiol S, Bogdanovic G, Buggert M, Ljunggren HG, Hober S, Nilsson P, Aleman S, Sallberg Chen M. Salivary IgG to SARS-CoV-2 indicates seroconversion and correlates to serum neutralization in mRNA-vaccinated immunocompromised individuals. Med. 2022 Feb 11;3(2):137-153.e3. doi: 10.1016/j.medj.2022.01.001. Epub 2022 Jan 20. PMID 35075450

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of the primary study population (immunosuppressed participants ) took place at Karolinska University Hospital.
  The control group was recruited, for example, from among staff at Karolinska University Hospital and, if necessary, from other healthcare units or facilities, such as primary care centers, via the Always Open app, recruitment flyers, or advertisements.
Pre-assignment Details: 781 participants were screened for the study at at Karolinska University Hospital between February 12th and 22nd, 2021 and 539 were included and recived the first vaccin dose. The main reasons for screening failure were previous COVID-19 infection, patient refusal, and that some study subjects already had been vaccinated outside the study.
Groups:
- All Immunocompromised Patients: This arm consists of individuals with a primary immunodeficiency disorder.
- Controls: The control group consisted of individuals without a primary immunodeficiency disorder.
Period: Overall Study
Arm/Group | All Immunocompromised Patients | Controls
Started | 449 | 90
Completed | 439 | 90
Not Completed | 10 | 0
Not completed — Adverse event, serious fatal | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Died in original disease | 2 | 0
Not completed — Leukemia relapse (more than 6 weeks after dose 2) | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | All Immunocompromised Patients | Controls | Total
Number analyzed (Participants) | 449 | 90 | 539
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 181 | 27 | 208
  >=65 years | 268 | 63 | 331
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 242 | 51 | 293
  Male | 207 | 39 | 246
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 449 | 90 | 539
Ongoing immunosuppression at baseline [Count of Participants; unit: Participants]
  Corticosteroids | 26 | 0 | 26
  Other immunosuppressive agents | 159 | 0 | 159
  No ongoing immunosuppression at baseline | 264 | 90 | 354
Immunogloublin G (IgG) level at baseline [Median (Full Range); unit: Immunglobulin G, IgG (g/L)] | 9.9 [1.0 to 34.4] | 11.0 [7.2 to 21.2] | 10.1 [1.0 to 34.4]
Absolute lymphocyte count(10^9 cells/L) at baseline [Median (Full Range); unit: Absolute lymphocyte count (10^9 cells/L)] | 1.6 [0.2 to 112.6] | 1.8 [1.0 to 4.1] | 1.6 [0.2 to 112.6]

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Seroconversion, Defined as Development of Immunoglobulin G (IgG) Antibodies Against Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) After Vaccination of 2 Doses in Seronegative Individuals.
Description: Proportion (95% confidence interval, CI) seroconverting to positive response to SARS-CoV-2 IgG serology test after two doses of vaccine, measured 2 weeks after second dose of vaccine.
Time Frame: 2 weeks after second dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | All Immunocompromised Patients | Controls
Number analyzed (Participants) | 388 | 78
Participants
  Seroconverted | 280 | 78
  Seronegative | 108 | 0
Statistical Analysis 1: Comparison: All Immunocompromised Patients vs Controls; Test type: Other; p < 0.05, Fisher Exact — The reported p-value was calculated

2. Secondary Outcome: Assessment of Any Adverse Events (AE) of the Given Vaccine.
Description: Proportion (95% CI) who experience adverse events, with AE/SAE/SUSAR (after dose 1)
Time Frame: Duration of 0-14 days after the first vaccine dose.
Measure: Count of Participants; unit: Participants
Arm/Group | All Immunocompromised Patients | Controls
Number analyzed (Participants) | 449 | 90
Participants
  AE | 94 | 6
  SAE | 10 | 0
  SUSAR | 1 | 0
  No AE/SAE/SUSAR | 344 | 84

3. Secondary Outcome: Assessment of Any Adverse Events (AE) of the Given Vaccine.
Description: Proportion (95% CI) who experience adverse events, with AE/SAE/SUSAR (after dose 2)
Time Frame: Duration of 0-14 days after the second vaccine dose.
Measure: Count of Participants; unit: Participants
Arm/Group | All Immunocompromised Patients | Controls
Number analyzed (Participants) | 446 | 88
Participants
  AE | 87 | 5
  SAE | 13 | 0
  SUSAR | 0 | 0
  No AE/SAE/SUSAR | 346 | 83

4. Secondary Outcome: Frequency Who Experience Local and Systemic Reactions
Description: Number and proportion (95% CI) who experience local and systemic reactions (after dose 1)
Time Frame: After the first vaccin dose
Measure: Count of Participants; unit: Participants
Arm/Group | All Immunocompromised Patients | Controls
Number analyzed (Participants) | 444 | 89
Participants
  Any reaction (grade 1 - 4) | 378 | 71
  No reaction | 66 | 18
Statistical Analysis 1: Comparison: All Immunocompromised Patients vs Controls; Test type: Other; p < 0.05, Chi-squared

5. Secondary Outcome: Frequency Who Experience Local and Systemic Reactions
Description: Number and proportion (95% CI) who experience local and systemic reactions (after dose 2)
Time Frame: After the second vaccin dose
Measure: Count of Participants; unit: Participants
Arm/Group | All Immunocompromised Patients | Controls
Number analyzed (Participants) | 422 | 87
Participants
  Any reaction (grade 1 - 4) | 337 | 74
  No reaction | 85 | 13
Statistical Analysis 1: Comparison: All Immunocompromised Patients vs Controls; Test type: Other; p < 0.05, Chi-squared

6. Secondary Outcome: Frequency of SARS-CoV-2 Infection Documented by PCR Test.
Description: Proportion (95% CI) diagnosed with a new SARS-CoV-2 infection confirmed by a positive PCR test
Time Frame: 0 - 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | All Immunocompromised Patients | Controls
Number analyzed (Participants) | 388 | 78
Participants
  Yes | 18 | 2
  No | 370 | 76

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded from the time of inclusion until visit 4, which occurred two weeks after administration of the second vaccine dose. Serious Adverse events (SAE) were documented up to visit 5, six weeks after the second vaccine dose.
Description: All Adverse Events (AE) were documented, exceptions included medical events that were anticipated sequelae of the underlying condition, such as exacerbation of the primary disease.
Groups:
- All Immunocompromised Patients: This arm consisted of individuals with a primary immunodeficiency disorder.
Arm/Group | All Immunocompromised Patients | Controls
All-Cause Mortality (participants affected / at risk) | 5/449 | 0/90
Serious Adverse Events (participants affected / at risk) | 23/449 | 0/90
Other Adverse Events (participants affected / at risk) | 173/449 | 11/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Immunocompromised Patients (N=449) | Controls (N=90)
Increased CRP (Investigations) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 2 (2) | 0 (0)
Surgery for colon carcinoma (Surgical and medical procedures) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Organ rejection (General disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increase/aspartate aminotransferase increase (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0)
Bone infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (3) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Immunocompromised Patients (N=449) | Controls (N=90)
Hypertension (Vascular disorders) | 13 (13) | 0 (0)
Superficial thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 3 (3) | 0 (0)
Lymph node punction (Surgical and medical procedures) | 1 (1) | 0 (0)
Increase thirst (General disorders) | 1 (1) | 0 (0)
Localized edema (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 2 (2) | 0 (0)
Fever (General disorders) | 2 (2) | 0 (0)
Vaccination site lymphadenopathy (General disorders) | 6 (6) | 1 (1)
Chest pain (General disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 10 (10) | 3 (3)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Unpleasantness while breathing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Development of bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Nightmares (Psychiatric disorders) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (4) | 0 (0)
Cholesterol high (Investigations) | 1 (1) | 0 (0)
Leukopenia (Investigations) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 17 (17) | 0 (0)
Pancytopenia (Investigations) | 2 (2) | 0 (0)
Monocyte count increased (Investigations) | 6 (6) | 0 (0)
Neutrophil count deceased (Investigations) | 5 (5) | 0 (0)
Increased lymphocyte count (Investigations) | 2 (2) | 0 (0)
Creatinine increased (Investigations) | 17 (17) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 4 (4) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 6 (6) | 0 (0)
Memory impairment (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Increased neutrophil count (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 7 (7) | 0 (0)
External otitis (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0)
Mucositis (Gastrointestinal disorders) | 4 (5) | 0 (0)
Increased LFTs (Hepatobiliary disorders) | 9 (9) | 0 (0)
Increased AST/ALT (Hepatobiliary disorders) | 11 (11) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin rash (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
GVHD (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Enlarged thyroid gland (Endocrine disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Traumatic knee injury (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Tendititis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Covid-19 (Infections and infestations) | 4 (4) | 2
Shingles (Infections and infestations) | 1 (1) | 0 (0)
BK-viremia (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis obliterans (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (6) | 0 (0)
Upper respiratory infection (Infections and infestations) | 21 (22) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0)
Strongyloides infection (Infections and infestations) | 1 (1) | 0 (0)
Bacterial infection UNS (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 3 (3) | 0 (0)
Cytomegalovirus infection reactivation (Infections and infestations) | 2 (2) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
GVHD in eye (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/59/NCT04780659/Prot_SAP_000.pdf